CLINICAL TRIAL: NCT03019874
Title: Observational Study With Mode of Action-Analysis of Cystorenal Cranberry Extract in Patients With Recurrent Urinary Tract Infections
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Other Study IDs: Cranberry
Record Dates: First submitted 2017-01-02; First posted 2017-01-13 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Dietary Supplement: Cranberry Extract — 3 x Cystorenal Cranberry plus daily for 6 months (contains 300 mg Cranberry-Extract, 100 mg Pumpkin seeds-Extract, 20 mg Vitamin C und 0,47 mg Riboflavin)

SUMMARY:
The main focus of this observational study is to analyze the possible effects of cranberry dietary supplements on the intestinal microbiota in women with recurrent uncomplicated urinary tract infections. In a secondary analysis the possible influence of the microbiota changes on the recurrence frequency in the follow-up should be analyzed.

ELIGIBILITY:
Inclusion criteria:

• chronic recurrent urinary tract infections (≥3 infections per year or 2 infections in the last 6 months)

Exclusion Criteria:

* renal insufficiency (GFR <60),
* anatomical or known structural causes of urinary tract infections
* regular consumption of probiotics or probiotic yogurts (at least 5x / week)
* intake of antibiotics in the last 4 weeks
* intake of Marcumar
* simultaneous participation in another study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic recurrent Urinary Tract Infections
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-01; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of urinary tract infections | In the 6-month prospective observation period compared to a 6-month retrospective period

SECONDARY OUTCOMES:
Quality of life (SF-36) | Baseline, 4 weeks, 8 weeks, 6 months

OTHER OUTCOMES:
Stool analysis: Intestinal microbiome by sequencing 16S rRNA | Baseline, 4 weeks, 8 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité University Medical Center
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany